CLINICAL TRIAL: NCT02060474
Title: Thyroid Hormone Analog Therapy of Patients With Severe Psychomotor Retardation Caused by Mutations in the MCT8 Thyroid Hormone Transporter: The Triac Trial.
Brief Title: Thyroid Hormone Analog Therapy in MCT8 Deficiency: Triac Trial Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, W. Edward Visser, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT8-2014-1; 2014-000178-20 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-12 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Allan-Herndon-Dudley Syndrome
Keywords: Allan-Herndon-Dudley Syndrome; MCT8; Triac; Therapeutic Trial
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — 3,3',5-triiodothyroacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AHDS patients (Experimental): all AHDS recruited for this study will be located in the experimental arm and will receive the investigational medicinal product Triac. The Triac dose will be individually titrated to the optimal dose level.
  Interventions: Drug: Triac

INTERVENTIONS:
Drug: Triac — Triac is a naturally occuring T3 metabolite with similar bioactivity and receptor binding profile.
  Other Names: Tiratricol, Téatrois, TA3

SUMMARY:
This therapeutical trial will be conducted in patients with the Allan-Herndon-Dudley Syndrome (AHDS), which is mutations in MCT8.

MCT8 is a thyroid hormone (TH) transporter which is crucial for the transport of TH from the blood into different tissues. Dysfunction of MCT8 results in a lack of TH (hypothyroidism) in tissues that depend on MCT8 for TH uptake. This local hypothyroidism in the brain of these patients causes severe psychomotor retardation.

In addition, TH serum parameters are highly abnormal in AHDS: high T3, low T4 and normal TSH levels. The high serum T3 levels cause local hyperthyroidism in tissues that do not depend on MCT8 for cellular transport of TH, resulting in a low body weight and reduced muscle mass.

Currently, no adequate treatment is available for the AHDS. A T3 analog that does not depend on MCT8 for its cellular entry could, at least partially, restore the abnormalities found in AHDS. Several in vivo, in vitro and animal studies have shown that the T3 analog Triac is a very promising candidate:

1. Triac binds to the same TH receptors as T3;
2. Cellular uptake of Triac does not depend on functional MCT8. Hence, in AHDS patients Triac will also be available in tissues that require functional MCT8 for TH uptake, e.g. the brain;
3. In vitro studies have shown that neuronal cells differentiate equally well in the presence of either Triac or T3;
4. In Mct8 deficient mice, Triac is taken up by the brain and suppresses serum TSH levels; consequently, serum T3 and T4 levels were lowered;
5. Triac is the treatment of choice in patient with the resistance to thyroid hormone (RTH) syndrome. Patient with RTH have high serum TSH and thyroid hormone levels, which shows strong similarities to the profile found in AHDS patients; the longstanding experience with Triac in RTH indicates its safety and tolerability .

Thus, Triac treatment could result in normalization of the abnormal serum TH values in AHDS patients. Furthermore, Triac could replace the function of T3 in tissues that depend on MCT8 for TH uptake (e.g. brain).

The current trial will investigate if Triac treatment in ADHS patients

1. reduces the toxic effects of the high T3 levels
2. restores the local TH deficiency in brain.

DETAILED DESCRIPTION:
All patients were treated with Triac (Téatrois tablets 350 microgram, Rare Thyroid Therapeutics) by individualized dose-escalation, following a pre-defined dose-escalation protocol. After the initial dose of Triac (350 microgram) was administered and no predefined dose-limiting toxicities were observed, the daily dose was increased progressively in 350 microgram steps, with a goal of attaining serum total T3 concentrations within the target range of 1·4-2·5 nmol per liter. The maintenance Triac dose was continued throughout the rest of the study period, but could be further adjusted according to the dose-escalation protocol if T3 concentrations were outside the target range during control visits.

Patients were assessed for study outcomes at baseline and 12 months after starting Triac administration. In the interval, patients were evaluated and screened for clinical and biochemical signs of hypothyroidism or hyperthyroidism, adverse events were recorded and adherence to therapy was assessed. All study procedures were specified in standard operating procedures, and were performed by well-trained investigators. Neuropsychological tests were conducted according to their manual. All biochemical measurements were performed in a central laboratory (Erasmus Medical Centre). To account for any interference of Triac in the measurement of serum T3 concentrations, conventional methods were employed to correct for cross-reactivity.

ELIGIBILITY:
Inclusion Criteria:

* clinically relevant mutation in the MCT8 gene, resulting in the clinical phenotype of AHDS.

Exclusion Criteria:

* Major illness or recent major surgery (within 4 weeks) unrelated to AHDS
* Patients who are participating in ongoing RCTs of therapeutic interventions (including clinical trials of investigational medicinal products);
* Known allergy to components in Triac tablets;
* Patients that have any contra-indication for Triac treatment.

Ages: 1 Day to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
serum T3 concentrations | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12, participants will be evaluated with an expected average of 6 weeks. For statistical analysis baseline and month 12 will be compared
  Serum T3 concentrations will be determined to assess the effect of Triac
serum free T4 concentrations | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12 participants will be evaluated with an expected average of 6 weeks. For statistical analysis baseline and month 12 will be compared
  Serum free T4 concentrations will be determined to assess the effect of Triac (co-primary end-point, supportive to changes in T3).
serum TSH concentrations | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12 participants will be evaluated with an expected average of 6 weeks. For statistical analysis baseline and month 12 will be compared
  Serum TSH concentrations will be determined to assess the effect of Triac (co-primary end-point, supportive to changes in T3).
serum total T4 concentrations | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12 participants will be evaluated with an expected average of 6 weeks. For statistical analysis baseline and month 12 will be compared
  Serum total T4 concentrations will be determined to assess the effect of Triac(co-primary end-point, supportive to changes in T3).
serum reverse T3 concentrations | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12 participants will be evaluated with an expected average of 6 weeks. For statistical analysis baseline and month 12 will be compared
  Serum reverse T3 concentrations will be determined to assess the effect of Triac(co-primary end-point, supportive to changes in T3).

SECONDARY OUTCOMES:
Heart rate | baseline and month 12 will be compared
  Heart rate will be measures with an ECG and 24 h ambulatory monitoring
serum sex-hormone binding globulin concentrations | baseline and month 12 will be compared
  serum sex-hormone binding globulin concentrations will be measured as a proxi-parameter for tissue thyroid hormone status in the liver.
Body weight | baseline and month 12 will be compared
  Body weight will be measured in kg
Blood pressure | baseline and month 12 will be compared
  Blood pressure will be measured in mmHg
serum total cholesterol concentrations | baseline and month 12 will be compared
  serum total cholesterol concentrations will be measured as a proxi-parameter for tissue TH status in the liver.
serum creatine kinase concentrations | baseline and month 12 will be compared
  serum creatine kinase concentrations will be measured as a proxi-parameter for tissue TH status in the muscles.

OTHER OUTCOMES:
Monitoring of adverse effects. | up to one year (= whole study period)
  Family members and caregivers of the included patients will be asked to report all adverse effects to one of the investigators.
A routine trans-thoracic cardiac ultrasound | 12 months
  the effects of Triac on the heart function will be measured using cardiac ultrasonography during the first visit (T0) and after 12 months (T12), reflecting the effect of Triac on the heart over a period of 1 year.
ECG | Participants will be evaluated with an expected average of 2 weeks during months 1-3 of the trial. During months 4-12 participants will be evaluated with an expected average of 6 weeks.
  The effect of Triac on the heart rhythm will be assessed with an ECG
Bone Mineral Density (total body) | Bone mineral density will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
  Bone mineral density of total body will be measured by DXA scan
Motor function, using the Gross Motor Function Measure | baseline and month 12 will be compared
  motor function will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
Cognitive function using the Bayley Scales of Infant Development III | baseline and month 12 will be compared
  cognitive function will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
Adaptive behavior by the Vineland adaptive behavior scale | baseline and month 12 will be compared
  adaptive behavior will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
Bone Mineral Density of ultradistal ulna | Bone mineral density will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
  Bone mineral density of ultradistal ulna will be measured by DXA scan
Bone Mineral Density of ultradistal radius | Bone mineral density will be measured during the first visit of the trial (T0) and after 12 months (T12) reflecting the effect of Triac over a 1 year period
  Bone mineral density of ultradistal radius will be measured by DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: W.E. Visser, dr,, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Groeneweg S, Peeters RP, Moran C, Stoupa A, Auriol F, Tonduti D, Dica A, Paone L, Rozenkova K, Malikova J, van der Walt A, de Coo IFM, McGowan A, Lyons G, Aarsen FK, Barca D, van Beynum IM, van der Knoop MM, Jansen J, Manshande M, Lunsing RJ, Nowak S, den Uil CA, Zillikens MC, Visser FE, Vrijmoeth P, de Wit MCY, Wolf NI, Zandstra A, Ambegaonkar G, Singh Y, de Rijke YB, Medici M, Bertini ES, Depoorter S, Lebl J, Cappa M, De Meirleir L, Krude H, Craiu D, Zibordi F, Oliver Petit I, Polak M, Chatterjee K, Visser TJ, Visser WE. Effectiveness and safety of the tri-iodothyronine analogue Triac in children and adults with MCT8 deficiency: an international, single-arm, open-label, phase 2 trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):695-706. doi: 10.1016/S2213-8587(19)30155-X. Epub 2019 Jul 31. PMID 31377265